CLINICAL TRIAL: NCT05509881
Title: Continuous Glucose Monitoring in Dialysis Patients to Overcome Dysglycemia Trial
Acronym: CONDOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Connie Rhee, Professor of Medicine, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1668
Record Dates: First submitted 2022-08-15; First posted 2022-08-22 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hemodialysis; Diabete Mellitus; Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous glucose monitoring (CGM) arm (Experimental): During the intervention period, patients in the CGM arm will undergo continuous real-time "unblinded" CGM using Dexcom CGM devices.
  Interventions: Device: Continuous glucose monitoring (CGM)
- Usual care arm (Active Comparator): During the intervention period, patients in the usual care arm will conduct self-monitored blood glucose (SMBG) at least 4 times/day. At Weeks 6 and 12 of the intervention period, usual care arm patients will also undergo 10-days of blinded CGM data collection.
  Interventions: Device: Usual care (Self-monitored blood glucose)

INTERVENTIONS:
Device: Continuous glucose monitoring (CGM) — Patients in the CGM arm will undergo continuous real-time "unblinded" CGM using Dexcom CGM devices.
  Arms: Continuous glucose monitoring (CGM) arm
Device: Usual care (Self-monitored blood glucose) — Patients in the usual care arm will conduct self-monitored blood glucose at least 4 times/day.
  Arms: Usual care arm

SUMMARY:
This randomized controlled trial will investigate whether use of continuous glucose monitoring (CGM) vs. usual care with self-monitored blood glucose 1) enhances glycemic control, 2) reduces hypoglycemia risk, and 3) improves quality of life, diabetes distress, and fear of hypoglycemia in hemodialysis patients with diabetes mellitus.

DETAILED DESCRIPTION:
This is a parallel, two-arm randomized controlled trial comparing real-time CGM using Dexcom devices vs. usual care (self-monitored blood glucose 4-times/day) among 122 in-center hemodialysis patients with diabetes mellitus over a 12-week period. Our primary objective will be to determine the effects of CGM vs. usual care on glycemic control, defined by percent (%) of time in target glucose range (70-180 mg/dl). Our main and exploratory secondary objectives will be to determine the effects of CGM on CGM-indices of hypoglycemia, blood-based glycemic markers (HbA1c, glycated albumin, fructosamine), and patient-reported outcomes (health-related quality of life, diabetes distress, hypoglycemia fear). We will also evaluate feasibility endpoints by measuring CGM compliance during the intervention period and success/ease of implementing CGM training sessions among patients.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Age ≥18 years old
* End-stage kidney disease status receiving in-center hemodialysis ≥4 weeks
* Type 1 or type 2 diabetes
* Actively performing self-monitored blood glucose (SMBG) testing for ≥4 weeks
* ≥70% compliance wearing continuous glucose monitoring (CGM) device during the pre-trial period

Exclusion Criteria:

* Inability to provide informed consent or comply with the study protocol
* Limited visual acuity
* Inability to wear CGM device
* Prior use of CGM
* Active pregnancy or planning a pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Percent (%) of time in target glucose range (70-180 mg/dl) | 12 weeks
  Ascertained by continous glucose monitoring

SECONDARY OUTCOMES:
Percent (%) of time spent in hypoglycemia (<70 mg/dl) | 12 weeks
  Ascertained by continous glucose monitoring
Percent (%) of time spent in relative hypoglycemia (<100 mg/dl) | 12 weeks
  Ascertained by continous glucose monitoring
Glycemic variability | 12 weeks
  Ascertained by continous glucose monitoring
Hemoglobin A1c level | 12 weeks
  Ascertained by blood test
Fructosamine level | 12 weeks
  Ascertained by blood test
Glycated albumin level | 12 weeks
  Ascertained by blood test
Short Form 36 Survey Physical Component Summary Score | 12 weeks
  Ascertained by Short Form 36 Survey; Minimum-Maximum range is 0-100; Higher scores indicate better health-related quality of life
Diabetes Distress Scale Survey Score | 12 weeks
  Ascertained by Diabetes Distress Scale Survey; Minimum-Maximum range is 1-6; Higher scores indicate higher states of distress
Hypoglycemia Fear | 12 weeks
  Ascertained by Hypoglycemia Fear Survey II

OTHER OUTCOMES:
Continuous glucose monitoring compliance during the intervention period | 12 weeks
  CGM compliance will be ascertained by two metrics; 1) wearing the CGM device ≥6 days/week, and 2) % of time CGM is active, which is an automatically captured/reported metric on the Dexcom G6 device
Participant feedback on continuous glucose monitoring training sessions | 12 weeks
  Survey graded on a 5-point Likert scale; participants' qualitative feedback

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rhee CM, Kalantar-Zadeh K, Tuttle KR. Novel approaches to hypoglycemia and burnt-out diabetes in chronic kidney disease. Curr Opin Nephrol Hypertens. 2022 Jan 1;31(1):72-81. doi: 10.1097/MNH.0000000000000756. PMID 34750332
- [Background] Narasaki Y, Park E, You AS, Daza A, Peralta RA, Guerrero Y, Novoa A, Amin AN, Nguyen DV, Price D, Kalantar-Zadeh K, Rhee CM. Continuous glucose monitoring in an end-stage renal disease patient with diabetes receiving hemodialysis. Semin Dial. 2021 Sep;34(5):388-393. doi: 10.1111/sdi.13009. Epub 2021 Aug 10. PMID 34378258
- [Background] Rhee CM, Kovesdy CP, Kalantar-Zadeh K. Glucose Homeostasis, Hypoglycemia, and the Burnt-Out Diabetes Phenomenon in Kidney Disease. Semin Nephrol. 2021 Mar;41(2):96-103. doi: 10.1016/j.semnephrol.2021.03.004. PMID 34140100
- [Background] Rhee CM, Kovesdy CP, You AS, Sim JJ, Soohoo M, Streja E, Molnar MZ, Amin AN, Abbott K, Nguyen DV, Kalantar-Zadeh K. Hypoglycemia-Related Hospitalizations and Mortality Among Patients With Diabetes Transitioning to Dialysis. Am J Kidney Dis. 2018 Nov;72(5):701-710. doi: 10.1053/j.ajkd.2018.04.022. Epub 2018 Jul 20. PMID 30037725
- [Background] Rhee CM, Kovesdy CP, Ravel VA, Streja E, Brunelli SM, Soohoo M, Sumida K, Molnar MZ, Brent GA, Nguyen DV, Kalantar-Zadeh K. Association of Glycemic Status During Progression of Chronic Kidney Disease With Early Dialysis Mortality in Patients With Diabetes. Diabetes Care. 2017 Aug;40(8):1050-1057. doi: 10.2337/dc17-0110. Epub 2017 Jun 7. PMID 28592525